CLINICAL TRIAL: NCT01713218
Title: Evaluation of Tumoral Perfusion Modification by Dynamic Imaging After Neoadjuvant Chemotherapy Combining Gemcitabine and a Hedgehog Inhibitor (Vismodegib) in Patients With Resectable Pancreatic Adenocarcinoma
Brief Title: Effect on Tumor Perfusion of a Chemotherapy Combining Gemcitabine and Vismodegib Before Surgery in Pancreatic Cancer
Acronym: NEOPACHI-001
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jean-Luc Van Laethem (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Jean-Luc Van Laethem, MD, PhD, Erasme University Hospital
Organization: Erasme University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-003516-31
Record Dates: First submitted 2012-10-17; First posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Pancreatic Adenocarcinoma Resectable
Keywords: Pancreas; Cancer; Hedgehog inhibitor; Neoadjuvant chemotherapy; Dynamic imaging
MeSH Terms: conditions — Neoplasms | interventions — Gemcitabine; HhAntag691; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine+Vismodegib (Experimental): Neoadjuvant chemotherapy combining gemcitabine and Vismodegib during 4 weeks before surgery
  Interventions: Drug: gemcitabine; Drug: Vismodegib; Procedure: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: gemcitabine — Administrated intravenously at a dose of 1000 mg/m2 over 30 minutes weekly, week 1 to 4
  Other Names: GEMZAR
Drug: Vismodegib — 150 mg capsule, oral, once daily
  Other Names: GDC-0449
Procedure: Neoadjuvant chemotherapy — Combination of gemcitabine and Vismodegib during a window interval (4 weeks) before surgery

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) has one of the worst prognoses of all human cancers and is considered as a sanctuary, resistant to most of the drugs used. Identification of new molecular targets involved in its pathogenesis is urgently needed and required both proper and innovative efficacy assessment.

This proof-of-concept trial is studying the "dynamic" tumor response after the administration of a short course (4 weeks) neoadjuvant combination of gemcitabine and a Hedgehog inhibitor (Vismodegib) before surgery in patients with operable pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is characterized by a high stromal density and is a hypoperfused tumor, precluding cytotoxics delivery to the epithelial tumoral compartment. There is thus a rationale for combining chemotherapy and antistromal drugs like Hedgehog inhibitors. Targeting the resectable primary tumor offers an appropriate setting to (1) evaluate and monitor early treatment effects on the tumor, (2) correlate dynamic imaging changes (perfusion and diffusion coefficient) to pre- and post-therapeutic tissue changes, (3) identify specific predictive biomarkers for the drugs used (i.e. gemcitabine transporters and Hedgehog pathway genes and proteins) and (4) assess if this early "dynamic and biomolecular response" can predict treatment benefit and patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histo(cyto)logically proven ductal pancreatic adenocarcinoma
* Resectable or potentially resectable tumor; resectability assessed during a multidisciplinary meeting with expert surgeon and radiologist
* First line chemotherapy
* Age > 18 years
* WHO performance status (PS) grade 0 or 1;
* Absolute neutrophil count > 1.5 x 10 9 / L, platelets > 100 x 10 9/ L, creatinine clearance (Cockcroft and Gault formula) > 60 ml/min, haemoglobin level > 10 g/dl (transfusions authorized), bilirubin<1.5 g/dl;
* Optimal biliary drainage;
* Women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation of who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative serum or urine pregnancy test prior to treatment. All WCBP, all sexually active male patients, and all partners of patients must agree to use adequate methods of birth control throughout the study;
* Signed written informed consent.

Exclusion Criteria:

* Locally advanced non resectable or metastatic pancreatic adenocarcinoma
* Previous anticancer therapy for the pancreatic adenocarcinoma
* Biliary obstruction without endoscopic biliary drainage
* Any contre-indication for surgery
* Prior malignancy (except non-melanoma skin cancer, and in situ carcinoma of the uterine cervix treated with a curative intent and any other tumor in complete remission with a disease-free interval > 3 years)
* Uncontrolled congestive heart failure or angina pectoris, myocardial infarction within 1 year prior to study entry, uncontrolled hypertension (systolic pressure > 160 mm or diastolic pressure > 100 mm under well conducted antihypertensive treatment), QT prolongation
* Major uncontrolled infection
* Severe hepatic impairment
* Any medical, psychological, or social condition, which, in the opinion of the investigator, could hamper patient's compliance to the study protocol and/or assessment/interpretation of the data
* Pregnant or lactating women, or patients of both genders with procreative potential not using adequate contraceptive methods
* Patients receiving or having received any investigational treatment within 4 weeks prior to study entry, or participating to another clinical study;Subject previously enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
"Dynamic" tumor response rate as defined by a 20% modification of tumoral perfusion and cellular density parameters. | 4 weeks (duration of the neoadjuvant chemotherapy).
  In order to detect changes in the tumor microenvironment and to monitor treatment efficacy, Dynamic Contrast-Enhanced-Magnetic Resonance Imaging (DCE-MRI) and Diffusion Weighted-Magnetic Resonance Imaging (DW-MRI) constitute tools more and more used. The acquired data can be analyzed using a pharmacokinetic model to obtain quantitative parameters relative to tissue perfusion and vascular permeability (Ktrans, a volume transfer constant of contrast agent between blood plasma and the extravascular extracellular space; Apparent Diffusion Coefficient as a surrogate marker of tissue cellularity). DCE/DW-MRI will be achieved weekly before each neoadjuvant chemotherapy treatment and before surgery. Each patient will be his/her own control by comparing serial imaging results with those of the baseline MRI.

SECONDARY OUTCOMES:
Number of participants with adverse events as assessed by National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Effects (CTCAE) V4.0. | End of study follow-up (up to 2 years).
  Number of participants with (serious) adverse events will be considered as a measure of safety of the whole therapeutic sequence (gemcitabine + Hedgehog inhibitor+ surgery).

OTHER OUTCOMES:
Tumor response as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. | 4 weeks (duration of the neoadjuvant chemotherapy).
Effect of treatment on selected biomarkers in tumor resection specimens. | 4 weeks (duration of the neoadjuvant chemotherapy).
  The objective is to identify within pre-therapeutic samples and surgical specimens several specific biomarkers involved (1) in the Hedgehog signalling pathway (GLI1, Sonic Hedgehog, Patched, Smoothened immunohistochemical patterns protein expression) and predicting response to anti-Hh therapy, (2) in the metabolization of gemcitabine (human equilibrative nucleoside transporter 1, deoxycytidine kinase) and predicting response to gemcitabine therapy, and (3) in the relative contribution of both anti-Hh therapy and gemcitabine therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Van Laethem, MD, PhD, Principal Investigator — Erasme University Hospital
Locations (2):
- Belgium (2):
  - Antwerp University Hospital (UZA), Edegem, Antwerpen
  - Erasme University Hospital (ULB), Brussels